CLINICAL TRIAL: NCT06849622
Title: Auto-antibody Dosage From Blood Spots for Diagnosis of Type 1 Diabetes and Celiace Disease
Acronym: CELDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CELDI
Record Dates: First submitted 2025-02-20; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Celiac Disease in Children; Diabetes Mellitus, Type I; Screening
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test on blood sample (diagnosis of celiac and diabetes disease) (Other)
  Interventions: Diagnostic Test: Test on blood sample
- test on dried blood spot (celiac and diabetes patients) (Other)
  Interventions: Diagnostic Test: Test on dried blood sample

INTERVENTIONS:
Diagnostic Test: Test on blood sample — The blood sample will be drawn by venipuncture during clinical routine. The serum will be tested for coeliac or diabetes 1 auto-antibodies, using Elisa test.
  Arms: Test on blood sample (diagnosis of celiac and diabetes disease)
Diagnostic Test: Test on dried blood sample — A finger prick will be used to collect Dried blood Spot (DBS) on a special card. The eluted blood spot will be tested, for coeliac and diabetes 1 auto-antibodies, using the same method used for serum, and the same cut-offs for positivity and negativity (Elisa tests)
  Arms: test on dried blood spot (celiac and diabetes patients)

SUMMARY:
Early diagnosis of type 1 diabetes and celiac disease is very useful, allows early therapy and prevents deaths from the onset of diabetic ketoacidosis. This is a pilot study on screening of autoantibodies of type 1 diabetes and celiac disease in tuscany patients. The study aims to evaluate the concordance between the screening results obtained using two different matrix (blood drop spots on card and serum) in the search for autoantibodies for celiac disease and for type 1 diabetes. Moreover, it will be evaluated the feasibility and acceptability of the screening on a sample of the population enrolled in the territory through the participation of pediatricians.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 2-13 years
* Patients with a confirmed diagnosis of type 1 diabetes or celiac disease (positive controls) and children who do not have type 1 diabetes or celiac disease or autoantibodies associated with these pathologies (controls)
* Obtained informed consent

Exclusion Criteria:

* none

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Comparability between spot and serum tests of the following parameters tissue transglutaminase Immunoglobuline A (tTg IgA) test, reference values <16 Units/ml | Baseline

SECONDARY OUTCOMES:
Comparability between spot and serum tests of the following parameters: anti-insulin antibodies (IAA) test, reference values <10 Units/ml | Baseline
Comparability between spot and serum tests of the following parameters: protein tyrosine phosphatase antibodies (IA2) test, reference values <7.5 Units/ml | Baseline
Comparability between spot and serum tests of the following parameter glutamic acid decarboxylase antibodies (GAD-65) test, reference values <5.5Units/ml | Baseline
Comparability between spot and serum tests of the following parameter zinc transporter 8 (ZnT8) test, reference values <15Units/ml | Baseline
Antibody titers (Units/ml) for coeliac disease autoantibodies and type 1 diabetes | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital IRCCS, Florence, Italy, Italy

IPD SHARING:
Plan to Share IPD: No